CLINICAL TRIAL: NCT03723421
Title: The Effect of the Rapid Injection Technique Without Aspiration on Pain Level in Intramuscular Vaccination- A Single-blind Randomized Controlled Trial
Brief Title: Rapid Injection Technique Without Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, İLKNUR GÖL, PhD RN, Asistant PROFESSOR, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/9
Record Dates: First submitted 2018-10-26; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Pain
Keywords: pain management; Vaccination; Aspiration
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As the study was a single-blind trial, the pain assessment was performed by another nurse, in the second minute after the injection, using the numerical pain rating scale, in order to provide neutrality. The nurse was informed by the researcher about the use of the scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid Injection Group Without Aspiration (Experimental): The tetanus vaccine was applied into the deltoid muscle of the left arm in the sitting position by rapid injection technique without aspiration.
  Interventions: Other: Rapid Injection Group Without Aspiration
- Control (Experimental): The tetanus vaccine was applied into the deltoid muscle of the left arm in the sitting position with the standard injection technique.
  Interventions: Other: Control

INTERVENTIONS:
Other: Rapid Injection Group Without Aspiration — After filling in the personal information form, the tetanus vaccine was administered by using rapid injection without aspiration technique (the injector was held at 90 degrees, it was pricked into tissue rapidly, and the drug was given in 1-2 seconds without performing aspiration). (the injector was held at 90 degrees, it was pricked into tissue rapidly, and the drug was given in 1-2 seconds without performing aspiration). 2 days after the vaccination, the researcher got in contact with the students in the intervention and the control groups in order to ask whether a local side effect developed in the vaccination site or not.
  Arms: Rapid Injection Group Without Aspiration
Other: Control — After filling in the personal information form, the tetanus vaccine was made in accordance with the standard injection technique included in the application (the injector was held at 90 degrees, it was pricked into tissue, and the drug was given in 5-10 seconds after performing aspiration). 2 days after the vaccination, the researcher got in contact with the students in the intervention and the control groups in order to ask whether a local side effect developed in the vaccination site or not.
  Arms: Control

SUMMARY:
This experimental, single-blind, randomized controlled trial study was conducted to compare the effect of the rapid injection technique without aspiration on pain level in the vaccination for the young adult students. The population of the study consisted of the nursing students who had to be tetanus vaccinated as a protective measure. The students were divided into two groups, as the rapid injection technique without aspiration and control group. The Numerical Rating Scale was used to determine the perceived pain level

DETAILED DESCRIPTION:
Study Design; This was an experimental, single-blind, randomized controlled trial.

Study Population and Study Sample; The study was conducted in Turkey, in a family health center (FHC) in Central Anatolia Region. The population of the study consisted of the nursing students (n:125) of the faculty of health sciences who had to be tetanus-vaccinated as a protective measure before the clinical practice. Sample selection was not performed in the study and the whole population was tried to be reached. However, as 53 students were vaccinated before and 2 students used a painkiller before the vaccination, the sample of the study consisted of a total of 70 students.

The distributions of the students, who came to the family health center for the vaccination and were in accordance with the inclusion criteria, to the intervention group in which the rapid injection technique without aspiration was applied and the control group in which no intervention were applied by the simple randomized method. The papers with the same color and folding shape that represented the two study groups were put into a cloth bag. In order to provide the randomized distribution and reduce all the negative effects, the required explanation was made to the individuals to be vaccinated and they were requested to pull a paper randomly from the bag. In this way, the groups were balanced and totally 35 students were included in each group.

The personal information form was filled for each individual, who came to the FHC for the vaccination and agreed to participate in the study, before the procedure. The tetanus vaccine was applied into the deltoid muscle of the left arm in the sitting position in both the intervention and the control groups in the vaccination room. All the vaccines were made by a single researcher in order to eliminate the vaccination differences.

Outcome Measures Pain Level; As the study was a single-blind trial, the pain assessment was performed by another nurse, in the second minute after the injection, using the numerical pain rating scale, in order to provide neutrality. The nurse was informed by the researcher about the use of the scale. The nurses had no conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* healthy students,
* who did not take any painkiller before the vaccination,
* agreed to participate in the study and gave verbal consent were included in the study.

Exclusion Criteria:

* the individuals with pain and/or acute pyretic disease,
* who underwent topical anesthesia and/or used any painkillers were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Pain severity | 2 MONTHS
  As the study was a single-blind trial, the pain assessment was performed by another nurse, in the second minute after the injection, using the numerical pain rating scale, in order to provide neutrality. The nurse was informed by the researcher about the use of the Numerical Pain Rating Scale (NPRS). NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes (Rodrigues, 2001; Hawker, 2011). The scale is composed of numbers between 0 and 10. The pain scoring is performed in the way that the individual chooses the closest point related to his/her pain. "0 point" signifies no pain and "10 points" signify worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin Univesity, Çankiri, Turkey (Türkiye)